CLINICAL TRIAL: NCT04067219
Title: Determinants of Skin, Muscle and Bone Aging in HIV-1 Infected Patients
Brief Title: SkIn, Muscle and Bone Aging Determinants in HIV Infected-patients.
Acronym: SIMBAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2011/02
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: HIV-1-infection; Marker; Structural
Keywords: Alterations
MeSH Terms: interventions — Absorptiometry, Photon; Weights and Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): HIV-1 infected patients
  Interventions: Procedure: DXA (dual-energy x-ray absorptiometric) measurement

INTERVENTIONS:
Procedure: DXA (dual-energy x-ray absorptiometric) measurement — DXA, evaluation of muscular function and muscle strength; neurocognitive tests; non invasive analysis of mechanical skin properties; food frequency questionnaire; laboratory assessment (25 hydroxy vitamin D, calcium/phosphate metabolism, bone remodelling markers, T cell activation).

SUMMARY:
this study consists of the study of markers of skin, muscular, neurocognitive and bone aging in HIV infected adults and to compare the frequency of these signs to the general population of same gender and age.

DETAILED DESCRIPTION:
Nowadays, the elevated frequency of cancers as well as cardiovascular, neurocognitive and bone diseases seems to denote a process of accelerated aging in the treated HIV-infected population of western countries, who are 40 to 50 years old in median. Markers of age-related alterations should be compared to the distribution among the general population whenever possible, to disentangle the effect of HIV and "normal" ageing or ageing due to other conditions. Common mechanisms should be better understood, more specifically those related to the impact of tobacco, antiretroviral treatments, and nutritional components. For markers of skin, muscle, neurocognitive function and bone ageing, the distribution of the general population is available and, in addition, alteration of these markers might have common mechanisms, such as insufficiency in 25 hydroxy vitamin D or nutritional parameters. Therefore, a joint study of these three organs seems particularly relevant.

This aim is to study markers of skin, muscular, neurocognitive and bone aging in HIV infected adults and to compare the frequency of these signs to the general population of same gender and age.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients included in the TISSOS-VIH substudy of the ARNS CO3 Aquitaine Cohort or who had a DXA measurement of the lumbar spine, femoral neck, and total body between 2004 and 2011 at the University Hospital of Bordeaux,
* > 18 years
* Affiliated to the medical insurance
* Having had at least one DXA measurement prior to the SIMBAD study visit
* Written informed consent for the SIMBAD study

Exclusion Criteria:

* Hepatitis C virus co-infection
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2012-05-03 (Actual); Primary Completion 2013-01-03 (Actual); Study Completion 2013-12-19 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an alteration in bone, muscle, neurocognitive or skin parameters | At the earliest at the inclusion visit and within a 9-month window after inclusion
  presence of osteoporosis or osteopenia on DXA (T-score < -2.5 and <-1, respectively), locomotor test results > 2 standard deviations of the mean of the general population, presence of premature hair whitening in patients aged < 40 years (defined by>50% of gray hair before the age of 40)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick MERCIE, Pr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No